CLINICAL TRIAL: NCT01432769
Title: Effect of Enteral Nutrition in the Outcome of Patients With Cardiovascular Surgery
Brief Title: Enteral Nutrition After Cardiovascular Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Lnca Krisein Alejandra Martinez Fuentes, DEGREE IN NUTRITION AND FOOD SCIENCE, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-1001-24
Record Dates: First submitted 2011-09-07; First posted 2011-09-13 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Malnutrition; Heart Disease
Keywords: enteral nutrition; malnutrition; cardiac surgery
MeSH Terms: conditions — Malnutrition; Heart Diseases | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- individualized diet (Active Comparator): patients will receive a diet individualized to their calorie and protein requirements besides to dietary supplementation with a polymeric formula
  Interventions: Dietary Supplement: dietary supplement high in energy and protein
- standardized diet (No Intervention): patients in the "standardized diet" will receive the dietary management established by the hospital

INTERVENTIONS:
Dietary Supplement: dietary supplement high in energy and protein — patients in the "standardized diet" will receive extra 500 kcal from the dietary supplement
  Other Names: Brand name: Supportan by Fresenius Kabi
  Arms: individualized diet

SUMMARY:
Effect of enteral nutrition in the outcome of patients has the objective to determine the effect of implementing a nutritional support protocol on the outcome of cardiovascular surgery patients, the main justification of the study its the prevalence of malnutrition over the hospitalized patients and the way this complication influence the treatment efficacy, the risk of complications over these patients, the costs, the prognosis, mortality and hospital stay.

This study will be a control clinical trial, randomized and double blind.

DETAILED DESCRIPTION:
INTRODUCTION: Malnutrition is a complication that occurs frequently in hospitalized patients and influencing treatment efficacy, risks of complications, costs, prognosis, mortality and hospital stay. Cardiac Cachexia is a complication that is characterized by weight loss and suggests different mechanisms to explain it: poor diet, intestinal malabsorption, impaired metabolism, loss of nutrients through the digestive tract or urinary tract, increased protein loss and decreased anabolism, increased basal metabolic rate. It is reported a reduction in mortality in cardiac patients with higher body mass index (BMI), this potential protective effect is known as the obesity paradox. In a clinical study to determine whether BMI influences the risk of mortality in acute decompensated heart failure, the authors compared the BMI of 108 927 hospitalized patients and noted that hospital mortality was decreased as BMI increased, decreasing the risk of death 10% for every 5 unit increase in BMI of patients. Moreover, the enteral nutrition within the first 48hr after surgery, helps maintain the integrity of the intestinal mucosa and reduces the secretion of catabolic hormones. A meta-analysis shows that 85% of high-risk surgical patients tolerate enteral nutrition in the early postoperative period. As a nutritional support in critically ill patients, enteral keeps physiological mechanisms, a lower incidence of complications and low cost. Nutritional support in critically ill patients has three objectives: to conserve body mass, modulate immune function and metabolic response to moderate stress.

OBJECTIVE OF THE STUDY: To determine the effect of implementing a nutritional support protocol on the outcome of cardiovascular surgery patients.

METHODOLOGY: The investigators performed a controlled clinical trial in adult patients, both genders admitted to the coronary intensive care UMAE. IMSS No.1, having undergone cardiac surgery with or without pump. There will be a nutritional screening and patients with malnutrition are included at random to group A (which will immunomodulatory individualized diet) or group B (conventional nutritional treatment). The protocol will be given nutritional support enterally during their hospital stay. The progress of nutritional status will be measured by weight, BMI, albumin, transferrin, total count of lymphocytes and total proteins in addition to the hospital stay, complications and mortality. A comparison of the effect of individualized nutritional support with a standard control group will be performed.

ANALYSIS: The results will be emptied in a database in Excel. The investigators will use statistical packages: NCSS 2007 (01/07/1919) and SPSS (15.0). Qualitative variables will be expressed as percentages, quantitative variables as mean and standard deviation if the distribution is normal. The results will be analyzed according to intention to treat. Comparison of nutritional status by various quantitative indicators will be made by paired t test or Mann Whitney according to their distribution. Categorical variables were expressed as proportions and compared using Chi Square test. All tests will be considered significant p values less than 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery for revascularization, valve implant.
* Patients with some degree of malnutrition or at risk of malnutrition according to the implementation of the Nutritional Risk Screening-2002.
* By letter of informed consent.

Exclusion Criteria:

* Patients with cancer diagnosis, liver disease, kidney disease.
* Patients who decide to come out the study
* Patients who are transferred to other hospitals
* Patients with complications that prevent them from receiving enteral nutritional.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-02 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
nutritional status | 15 days
  Will be monitoring anthropometric indicators of nutritional status: weight and BMI, during hospitalization and weekly basis. Will be monitoring the biochemical indicators of nutritional status, albumin, transferrin, total lymphocyte count and total protein during hospitalization and weekly basis.
  Will be monitoring dietary indicators of nutritional status, daily protein intake and total calories during the hospitalization and daily newspaper.

SECONDARY OUTCOMES:
Days of hospitalization | 15 days
  To measure the clinical course of patients will be reported the numbers of days of hospitalization of patients
Infectious complications | 15 days
  as a secondary objective of the research it will be a recorded the number of patients with infectious complications during hospitalization
Mortality | 15 days
  as a secondary objective of the research it will be a recorded the all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: sergio e solorio meza, Doctor, Study Director — Instituto Mexicano del Seguro Social; guadalupe reynaga ornelas, researcher, Study Chair — Guanajuato's University; krisein a martinez fuentes, Nutritionist, Principal Investigator — Secretary of Health
Locations (1):
- Mexican Institute of social security: highly specialized medical unit number 1 Bajio, León, Guanajuato, Mexico